CLINICAL TRIAL: NCT05437692
Title: A Prospective, Single Arm, Phase II Clinical Study on the Treatment of Locally Advanced Cervical Cancer (Ⅱ B to Ⅳ a) With Zimberelimab Combined With Concurrent Radiotherapy and Chemotherapy
Brief Title: Zimberelimab Combined With Concurrent Radiotherapy and Chemotherapy for Locally Advanced Cervical Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2022-213R
Record Dates: First submitted 2022-06-24; First posted 2022-06-29 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-06

CONDITIONS: Locally Advanced Cervical Cancer
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- zimberelimab plus concurrent radiotherapy and chemotherapy (Experimental): 19 patients will treated with zimberelimab plus concurrent radiotherapy and chemotherapy
  Interventions: Drug: zimberelimab combined With concurrent radiotherapy and chemotherapy

INTERVENTIONS:
Drug: zimberelimab combined With concurrent radiotherapy and chemotherapy — zimberelimab: 240 mg Q2W Intravenous drip，The maximum duration of medication shall not exceed one years; chemotherapy: Starting from the first week of radiotherapy and chemotherapy, cisplatin 40mg/m2 and paclitaxel 35mg/m2 were given intravenously for 30-60min; Radiotherapy: intensity modulated radiation therapy (IMRT) was used for external irradiation. The total dose of pelvic cavity and lymph drainage planning target area (PTV) was 45-50 gy/25-28f. The metastatic lymph nodes should be able to supplement or synchronously push 10-15 Gy; The internal irradiation was started within 2 weeks after the end of external irradiation treatment. The image-guided three-dimensional brachytherapy was used, and 30-40gy was added to make the total dose of point a reach 80-85 Gy, twice a week, 5-6gy each time. All radiotherapy was completed within 8 weeks.
  Other Names: GSL-010

SUMMARY:
This is a prospective, single arm, phase II clinical study on the treatment of locally advanced cervical cancer (Ⅱ B to Ⅳ a) with Zimberelimab combined with concurrent radiotherapy and chemotherapy.

DETAILED DESCRIPTION:
This study will include 19 patients with locally advanced cervical cancer to explore the efficacy and safety of Zimberelimab in combination with concurrent radiotherapy for them.

ELIGIBILITY:
Inclusion Criteria:

* FIGO 2018 stage IIB to IVA cervical cancer;
* Cervical squamous cell carcinoma, cervical adenocarcinoma or cervical adenosquamous carcinoma confirmed by histology;
* Have not received any radiotherapy for cervical cancer in the past, and have not received immunotherapy;
* Have measurable lesions (according to RECIST v1.1 standard);
* ECOG score: 0 ~ 1;
* 18~75 years old (calculated on the day of signing the informed consent);
* The estimated survival period exceeds 6 months;
* Before enrollment, try to provide enough tumor tissue samples (archived or fresh biopsy samples) to evaluate and confirm the expression of PD-L1 and to detect other biomarkers; Considering the accessibility of clinical specimens, there is no mandatory requirement for specimens;
* Women of childbearing age should agree to use contraceptives (such as intrauterine devices, contraceptives or condoms) during the study period and within ● months after the end of the study; Within 7 days before the study was enrolled, the serum or urine pregnancy test was negative, and must be non lactating patients;
* For the full organ function defined in the protocol, the test samples must be collected within 7 days before the start of the study treatment;
* The patients volunteered to join the study and signed the informed consent form.

Exclusion Criteria:

* The subjects have other histological subtypes except those permitted by inclusion criteria 2;
* Bilateral hydronephrosis, unless at least one side has been implanted with a stent or solved by a positioned nephrostomy;
* Those who are allergic to gadolinium, a common non-ionic CT contrast agent and a magnetic resonance contrast agent
* Have anatomical structure or tumor geometry or any other reasons or contraindications that cannot be treated with intracavitary brachytherapy or intracavitary and implantable brachytherapy;
* Severe hypersensitivity (≥ grade 3) to cepalimumab and / or any of its excipients;
* Participated in or had participated in clinical trials within 4 weeks before randomization;
* Have been vaccinated or will be vaccinated with live vaccine within 30 days before the first study treatment;
* Have received systemic immune stimulant, colony stimulating factor, interferon, interleukin and vaccine combination treatment within 6 weeks or 5 half lives (whichever is shorter) before the first administration;
* Within 7 days before the first administration, the patient has been diagnosed with immune deficiency or is receiving chronic systemic steroid therapy (the dose exceeds 10mg prednisone equivalent per day) or any other form of immunosuppressive therapy;
* Active autoimmune diseases requiring systemic treatment during the past two years (such as the use of disease regulating drugs, corticosteroids or immunosuppressive drugs);
* Have a history of (non infectious) pneumonia requiring steroid treatment or currently have (non infectious) pneumonia;
* Active infection requiring systematic treatment;
* Known HIV infection history;
* Known hepatitis B (defined as HBsAg reactivity) or known active hepatitis C virus (defined as detection of HCV RNA [qualitative]) infection history;
* Known history of active tuberculosis (TB; Mycobacterium tuberculosis);
* Received allogeneic tissue / solid organ transplantation;
* Central nervous system metastasis such as tumor brain metastasis;
* Patients with uncontrolled hydrothorax and ascites;
* Patients with movement disorders such as pathological fractures caused by tumor bone metastasis;
* Insufficient hematopoietic function of bone marrow (without blood transfusion within 14 days):
* Abnormal liver:
* Abnormal kidney:
* Risk of bleeding:
* Cardiovascular and cerebrovascular abnormalities:

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
ORR | one year
  Objective response rate based on RECIST v1.1

SECONDARY OUTCOMES:
adverse events | two years
  adverse events evaluation based on NCI-CTCAE 5.0
DCR | one year
  Disease control rate evaluation based on RECIST v1.1
OS | three years
  overall survival time
PFS | two years
  Progression free survival time

CONTACTS AND LOCATIONS:
Overall Officials: Lin Genlai, MD, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Shanghai Zhongshan hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared.

REFERENCES:
- [Result] Wright JD, Matsuo K, Huang Y, Tergas AI, Hou JY, Khoury-Collado F, St Clair CM, Ananth CV, Neugut AI, Hershman DL. Prognostic Performance of the 2018 International Federation of Gynecology and Obstetrics Cervical Cancer Staging Guidelines. Obstet Gynecol. 2019 Jul;134(1):49-57. doi: 10.1097/AOG.0000000000003311. PMID 31188324
- [Result] Arbyn M, Weiderpass E, Bruni L, de Sanjose S, Saraiya M, Ferlay J, Bray F. Estimates of incidence and mortality of cervical cancer in 2018: a worldwide analysis. Lancet Glob Health. 2020 Feb;8(2):e191-e203. doi: 10.1016/S2214-109X(19)30482-6. Epub 2019 Dec 4. PMID 31812369
- [Result] Koh WJ, Abu-Rustum NR, Bean S, Bradley K, Campos SM, Cho KR, Chon HS, Chu C, Clark R, Cohn D, Crispens MA, Damast S, Dorigo O, Eifel PJ, Fisher CM, Frederick P, Gaffney DK, Han E, Huh WK, Lurain JR, Mariani A, Mutch D, Nagel C, Nekhlyudov L, Fader AN, Remmenga SW, Reynolds RK, Tillmanns T, Ueda S, Wyse E, Yashar CM, McMillian NR, Scavone JL. Cervical Cancer, Version 3.2019, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2019 Jan;17(1):64-84. doi: 10.6004/jnccn.2019.0001. PMID 30659131
- [Result] Kokka F, Bryant A, Brockbank E, Powell M, Oram D. Hysterectomy with radiotherapy or chemotherapy or both for women with locally advanced cervical cancer. Cochrane Database Syst Rev. 2015 Apr 7;(4):CD010260. doi: 10.1002/14651858.CD010260.pub2. PMID 25847525
- [Result] Pakish JB, Jazaeri AA. Immunotherapy in Gynecologic Cancers: Are We There Yet? Curr Treat Options Oncol. 2017 Aug 24;18(10):59. doi: 10.1007/s11864-017-0504-y. PMID 28840453
- [Result] Mandal R, Chan TA. Personalized Oncology Meets Immunology: The Path toward Precision Immunotherapy. Cancer Discov. 2016 Jul;6(7):703-13. doi: 10.1158/2159-8290.CD-16-0146. Epub 2016 Apr 22. PMID 27107038
- [Result] Bonneville R, Krook MA, Kautto EA, Miya J, Wing MR, Chen HZ, Reeser JW, Yu L, Roychowdhury S. Landscape of Microsatellite Instability Across 39 Cancer Types. JCO Precis Oncol. 2017;2017:PO.17.00073. doi: 10.1200/PO.17.00073. Epub 2017 Oct 3. PMID 29850653
- [Result] Shao C, Li G, Huang L, Pruitt S, Castellanos E, Frampton G, Carson KR, Snow T, Singal G, Fabrizio D, Alexander BM, Jin F, Zhou W. Prevalence of High Tumor Mutational Burden and Association With Survival in Patients With Less Common Solid Tumors. JAMA Netw Open. 2020 Oct 1;3(10):e2025109. doi: 10.1001/jamanetworkopen.2020.25109. PMID 33119110
- [Result] Liu Y, Wu L, Tong R, Yang F, Yin L, Li M, You L, Xue J, Lu Y. PD-1/PD-L1 Inhibitors in Cervical Cancer. Front Pharmacol. 2019 Feb 1;10:65. doi: 10.3389/fphar.2019.00065. eCollection 2019. PMID 30774597
- [Result] Frenel JS, Le Tourneau C, O'Neil B, Ott PA, Piha-Paul SA, Gomez-Roca C, van Brummelen EMJ, Rugo HS, Thomas S, Saraf S, Rangwala R, Varga A. Safety and Efficacy of Pembrolizumab in Advanced, Programmed Death Ligand 1-Positive Cervical Cancer: Results From the Phase Ib KEYNOTE-028 Trial. J Clin Oncol. 2017 Dec 20;35(36):4035-4041. doi: 10.1200/JCO.2017.74.5471. Epub 2017 Nov 2. PMID 29095678
- [Result] Chung HC, Ros W, Delord JP, Perets R, Italiano A, Shapira-Frommer R, Manzuk L, Piha-Paul SA, Xu L, Zeigenfuss S, Pruitt SK, Leary A. Efficacy and Safety of Pembrolizumab in Previously Treated Advanced Cervical Cancer: Results From the Phase II KEYNOTE-158 Study. J Clin Oncol. 2019 Jun 10;37(17):1470-1478. doi: 10.1200/JCO.18.01265. Epub 2019 Apr 3. PMID 30943124
- [Result] Tamura K, Hasegawa K, Katsumata N, Matsumoto K, Mukai H, Takahashi S, Nomura H, Minami H. Efficacy and safety of nivolumab in Japanese patients with uterine cervical cancer, uterine corpus cancer, or soft tissue sarcoma: Multicenter, open-label phase 2 trial. Cancer Sci. 2019 Sep;110(9):2894-2904. doi: 10.1111/cas.14148. Epub 2019 Sep 3. PMID 31348579
- [Result] Naumann RW, Hollebecque A, Meyer T, Devlin MJ, Oaknin A, Kerger J, Lopez-Picazo JM, Machiels JP, Delord JP, Evans TRJ, Boni V, Calvo E, Topalian SL, Chen T, Soumaoro I, Li B, Gu J, Zwirtes R, Moore KN. Safety and Efficacy of Nivolumab Monotherapy in Recurrent or Metastatic Cervical, Vaginal, or Vulvar Carcinoma: Results From the Phase I/II CheckMate 358 Trial. J Clin Oncol. 2019 Nov 1;37(31):2825-2834. doi: 10.1200/JCO.19.00739. Epub 2019 Sep 5. PMID 31487218
- [Result] Santin AD, Deng W, Frumovitz M, Buza N, Bellone S, Huh W, Khleif S, Lankes HA, Ratner ES, O'Cearbhaill RE, Jazaeri AA, Birrer M. Phase II evaluation of nivolumab in the treatment of persistent or recurrent cervical cancer (NCT02257528/NRG-GY002). Gynecol Oncol. 2020 Apr;157(1):161-166. doi: 10.1016/j.ygyno.2019.12.034. Epub 2020 Jan 7. PMID 31924334
- [Result] Colombo N, Dubot C, Lorusso D, Caceres MV, Hasegawa K, Shapira-Frommer R, Tewari KS, Salman P, Hoyos Usta E, Yanez E, Gumus M, Olivera Hurtado de Mendoza M, Samouelian V, Castonguay V, Arkhipov A, Toker S, Li K, Keefe SM, Monk BJ; KEYNOTE-826 Investigators. Pembrolizumab for Persistent, Recurrent, or Metastatic Cervical Cancer. N Engl J Med. 2021 Nov 11;385(20):1856-1867. doi: 10.1056/NEJMoa2112435. Epub 2021 Sep 18. PMID 34534429
- [Result] Menderes G, Black J, Schwab CL, Santin AD. Immunotherapy and targeted therapy for cervical cancer: an update. Expert Rev Anticancer Ther. 2016;16(1):83-98. doi: 10.1586/14737140.2016.1121108. Epub 2015 Dec 7. PMID 26568261
- [Result] Wang CC, Chou HH, Yang LY, Lin H, Liou WS, Tseng CW, Liu FY, Liou JD, Huang KG, Huang HJ, Huang EY, Chen CH, Chang TC, Chang CJ, Hong JH, Lai CH. A randomized trial comparing concurrent chemoradiotherapy with single-agent cisplatin versus cisplatin plus gemcitabine in patients with advanced cervical cancer: An Asian Gynecologic Oncology Group study. Gynecol Oncol. 2015 Jun;137(3):462-7. doi: 10.1016/j.ygyno.2015.03.046. Epub 2015 Mar 28. PMID 25827291
- [Result] Thakur P, Seam R, Gupta M, Gupta M. Prospective randomized study comparing concomitant chemoradiotherapy using weekly cisplatin & paclitaxel versus weekly cisplatin in locally advanced carcinoma cervix. Ann Transl Med. 2016 Feb;4(3):48. doi: 10.3978/j.issn.2305-5839.2015.11.19. PMID 26904570

DOCUMENTS (1):
  • Informed Consent Form (2022-05-05): https://cdn.clinicaltrials.gov/large-docs/92/NCT05437692/ICF_000.pdf